CLINICAL TRIAL: NCT00465153
Title: The Combined Effects of Resistance Training and Flax Oil Supplementation Upon Inflammation in Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Gatorade Sports and Science Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bio-REB 06-211
Record Dates: First submitted 2007-04-20; First posted 2007-04-24 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Inflammation; Sarcopenia
Keywords: Inflammation; cytokines; sarcopenia; strength; muscle; aging; exercise
MeSH Terms: conditions — Inflammation; Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Flax oil
  Interventions: Dietary Supplement: flax oil containing alpha linolenic acid; Behavioral: Resistance exercise training
- 2 (Placebo Comparator): corn oil
  Interventions: Dietary Supplement: flax oil containing alpha linolenic acid

INTERVENTIONS:
Dietary Supplement: flax oil containing alpha linolenic acid — 14g alpha linolenic acid per day
  Other Names: WN Pharmaceuticals
Behavioral: Resistance exercise training — Resistance training
  Arms: 1

SUMMARY:
Loss of muscle mass and functional ability is a major concern for older individuals. Aging is associated with increased inflammation caused by release of hormone-like compounds termed "cytokines" which are involved in muscle protein degradation. Diets rich in ω-3 fatty acids decrease the production of pro-inflammatory cytokines, possibly by inhibiting production of lipids involved in cytokine synthesis. Our purpose is to assess the effect of dietary supplementation with an ω-3 fatty acid, α-linolenic acid (ALA) commonly found in flaxseed, combined with resistance training on pro-inflammatory cytokines, strength, and muscle mass in older adults. Progressive resistance training is considered to be the standard for increasing strength and muscle mass in older adults. We hypothesize that combining the two interventions will improve strength and muscle mass more than resistance training alone by modulating the inflammatory process associated with aging. Our proposed research will compare older individuals supplementing with ALA and placebo during a resistance training program.

DETAILED DESCRIPTION:
The specific aim is to determine the effect of progressive resistance training and α-linolenic acid supplementation for decreasing markers of inflammation and improving muscle mass and strength in older adults. This will be done by comparing older adults who will participate in the same resistance training program while supplementing their diet with either α-linolenic acid or placebo.

The hypotheses of this research are:

Resistance training combined with α-linolenic acid supplementation will decrease the pro-inflammatory cytokines interleukin-6 (IL-6) and tumour necrosis factor alpha (TNF-α), and increase strength and muscle mass more than resistance training and placebo supplementation in older individuals.

Sixty untrained males and females over 60 years of age will be recruited by newspaper ads. Subjects will be matched for sex and age and randomly assigned to supplement with 15 g/day α-linolenic acid (ALA) from flaxseed oil or placebo (corn oil) while participating in resistance training, 3 times per week for 12 weeks. The 15 g dose was chosen because it was effective for reducing pro-inflammatory cytokines in healthy adults over 4 weeks (Caughey et al., 1996). Twelve weeks of resistance training was chosen because it is effective for increasing muscle mass and strength in older adults (Chrusch et al., 2001). Our sample size of 30 subjects per group will be sufficient for detecting the expected changes in cytokines (Caughey et al., 1996) with a power of 80% and alpha level of 0.05. The primary dependent variables will be the pro-inflammatory cytokines IL-6 and TNF-α. Secondary dependent variables are chest press and leg press strength, lean tissue mass, and muscle thickness. A 2 (groups) x 2 (time, baseline and 12 weeks) ANOVA with repeated measures on the 2nd factor, will be used for analyses with alpha level of 0.05.

Methodology: Exercise Training: The exercise training will consist of a progressive resistance training program designed to increase skeletal muscle hypertrophy by having participants complete 12 different machine-based resistance exercises. The exercises will include: chest press, shoulder press, lat pulldown, bicep curl, triceps extension, leg press, knee flexion, knee extension, hip flexion/extension, and hip abduction/adduction. The subjects will complete between 3-4 sets of 6-12 repetitions at intensities between 65-80% of their 1 repetition maximum in a progressively overloaded fashion.

Biochemical Measures: Assessment of markers of inflammation will be done by biochemical blood analysis at baseline and after 12 weeks supplementation combined with resistance training. Blood will be drawn after an overnight night fast in the morning to account for changes due to diurnal variation. Approximately 10 mL of blood will be drawn from the antecubital vein of the arm. Serum will be assessed for the pro-inflammatory cytokines interleukin-6 and tumor necrosis factor-alpha using ELISA.

Fitness Testing: One repetition maximum (RM) strength tests will be done using chest press and leg press at baseline and 12 weeks. Subjects will complete a standardized warm-up of cycling and stretching before the strength test. The testing protocol will allow subjects to become familiar with the movement patterns of the resistance training machines before initiating the strength testing trials. Subjects will be gradually progressed to the maximal load that they can lift for the chest press and leg press. Once the subject is unable to complete a full repetition, the last successful attempt will be recorded as their 1RM.

Body Composition: Lean tissue and fat mass will be assessed by dual energy X-ray absorptiometry, and muscle thickness of the extensors and flexors of the elbows and knees will be determined by ultrasound at baseline and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 60y

Exclusion Criteria:

* allergies to flax or corn oil
* Smokers
* Consume more than 2 portions of oily fish per week
* Take prescription or over the counter medication or natural health products that are anti-inflammatory in nature
* Autoimmune or inflammatory disease
* Susceptible to bowel irritation
* Involved in resistance training equal to or greater than 1 time per week

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 and tumor necrosis factor-alpha at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Bench press and leg press strength, lean tissue mass, and muscle thickness of arm and leg flexors and extensors at 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan; Lisa Paus-Jenssen, M.D., Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada